CLINICAL TRIAL: NCT03716791
Title: The Effect of Methylsulfonylmethane (MSM) on Cardiometabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lindsey Miller (Other)
Responsible Party: Sponsor-Investigator, Lindsey Miller, Assistant Professor, Washington State University
Organization: Washington State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 16970-001
Record Dates: First submitted 2018-10-18; First posted 2018-10-23 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — dimethyl sulfone

STUDY DESIGN:
Intervention Model Description: Double-blind placebo controlled randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Control Group (Placebo Comparator): pill capsules containing white rice flour
  Interventions: Dietary Supplement: placebo
- Methylsulfonylmethane Group (Active Comparator): pill capsules containing MSM
  Interventions: Dietary Supplement: methylsulfonylmethane

INTERVENTIONS:
Dietary Supplement: methylsulfonylmethane — 3g per day
  Other Names: MSM
  Arms: Methylsulfonylmethane Group
Dietary Supplement: placebo — white rice flour
  Arms: Placebo Control Group

SUMMARY:
Obesity- related diseases are linked to elevated levels of inflammation, oxidative stress, and metabolic dysfunction. Methylsulfonylmethane (MSM) is a naturally occurring compound that demonstrates antioxidant and anti-inflammatory effects. Improvements in measures of metabolic health have been observed in mouse models of obesity and type 2 diabetes following MSM treatment. However, the effect of MSM on obesity-related risk factors for disease in humans has not been investigated. Therefore, the purpose of this investigation will be to determine whether MSM supplementation improves metabolic health, and markers of inflammation and oxidative status.

ELIGIBILITY:
Inclusion Criteria:

* overweight or obese adults without any diagnosed disease or current medications other than birth control. Participants must agree to maintain diet and physical activity levels throughout study.

Exclusion Criteria:

* normal weight adults, or overweight/obese adults that do not meet the criteria for metabolically unhealthy obesity. Individuals currently on medications, or with diagnosed disease. Pregnant or nursing women, or women planning to become pregnant within the study timeframe. Lack of access to reliable transportation to study site, lack of internet access, or non-english speaking.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-08-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline blood glucose at 4, 8, and 16 weeks | 0,4,8,16 weeks
Change from baseline blood cholesterol at 4, 8, and 16 weeks | 0,4,8,16 weeks
Change from baseline blood pressure at 4, 8, and 16 weeks | 0,4,8,16 weeks

SECONDARY OUTCOMES:
Change from baseline insulin at 4, 8, and 16 weeks | 0,4,8,16 weeks
Change from baseline resting metabolic rate at 16 weeks | 0 and 16 weeks
Change from baseline percent body fat at 4, 8, and 16 weeks | 0,4,8,16 weeks
Change from baseline in waist circumference at 4, 8, and 16 weeks | 0,4,8,16 weeks
Change from baseline in blood markers of inflammation and oxidative stress at 4, 8, and 16 weeks | 0,4,8,16 weeks
  Inflammatory markers will include c-reactive protein, interleukin-6, and Tumor necrosis factor-alpha. Oxidative stress will be determined by total antioxidant capacity assay.
Change from baseline in pulmonary function tests | 0, 4, 8, 16 weeks
  Pulmonary function tests include forced expiratory volume in 1 second to forced vital capacity ration and slow vital capacity measurement. Expired nitric oxide has also been included as a marker of pulmonary inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey E Miller, Ph.D, Principal Investigator — Washington State University
Locations (1):
- Washington State University, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No